CLINICAL TRIAL: NCT01806987
Title: A Randomized Efficacy Trial of the Kids in Transition to School (KITS) Program to Improve School Readiness of Children in Disadvantaged Communities
Brief Title: A Test of the Kids in Transition to School (KITS) Program in Disadvantaged Neighborhoods
Acronym: KITS-PN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine C. Pears, Senior Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R305A120391; R305A120391 (Other Grant/Funding Number: IES)
Record Dates: First submitted 2013-03-01; First posted 2013-03-08 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: School Readiness
Keywords: school readiness; literacy; social emotional skills; self regulation; caregiver involvement; socioeconomic disadvantage
MeSH Terms: conditions — Literacy; Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KITS Program (Experimental): The KITS Program consists of: (a) child school readiness play groups to facilitate the development of self-regulatory, social, and early literacy skills (2 times per week in summer, 1 time per week in the fall); and (b) a 12 session psychoeducational workshop to promote parent involvement in the child's early literacy and schooling and the use of effective parenting techniques (once per week in summer, bi-weekly in the fall).
  Interventions: Behavioral: KITS Program
- Services as usual (No Intervention): These include any services that the child and family might already be receiving in the community.

INTERVENTIONS:
Behavioral: KITS Program — The KITS Program is a 4-month psychosocial intervention for children at high risk for school difficulties and their caregivers. The intervention begins in the summer before kindergarten and continues across the first two months of kindergarten. The KITS intervention consists of: (a) child school readiness play groups to facilitate the development of self-regulatory, social, and early literacy skills (2 times per week in summer, 1 time per week in the fall); and (b) a 12 session psychoeducational workshop to promote parent involvement in the child's early literacy and schooling and the use of effective parenting techniques (once per week in summer, bi-weekly in the fall).
  Other Names: Kids in Transition to School Program
  Arms: KITS Program

SUMMARY:
The purpose of this project to determine whether the KITS Program, an intervention to improve early literacy, prosocial and emotion and behavior regulation domains of school readiness, improves school readiness and school outcomes in children from socioeconomically disadvantaged neighborhoods.

DETAILED DESCRIPTION:
PURPOSE: This project is a randomized efficacy trial of the KITS Program, an intervention to improve early literacy, prosocial and emotion and behavior regulation domains of school readiness, with children from socioeconomically disadvantaged neighborhoods. The project will extend the evidence on the efficacy of the intervention from two previous randomized efficacy trials of the KITS Program with special needs populations to examine the impacts of the intervention on the broader population of children from disadvantaged backgrounds in general education.

SETTING: The intervention will be conducted in elementary school classrooms in high-poverty, high-crime neighborhoods in a medium-sized metropolitan area of the Pacific Northwest during the summer before and the first 2 months of kindergarten.

POPULATION: This study involves the recruitment of 240 children who will be entering kindergarten in the fall and their families in three yearly cohorts (n = 80). The children will be recruited from neighborhoods that have been selected as some of the most disadvantaged in the state in terms of income and school readiness indicators.

INTERVENTION: The KITS Program is a high-intensity, short-term program timed to occur during the transition to kindergarten-a critical developmental milestone with far-reaching effects on school outcomes. The curriculum focuses on the early literacy, social, and self-regulation skills critical for success in kindergarten and on contextual characteristics (i.e., parent involvement in early literacy and positive parenting). KITS features 24 curriculum-based therapeutic playgroups focused on early literacy, social, and self-regulatory skills and 12 psychoeducational parent workshops focused on parent involvement in early literacy and positive parenting practices.

CONTROL CONDITION: The children in the services-as-usual condition will receive any early childhood learning services that they would typically receive prior to school entry. Services received will be assessed at each data time point.

RESEARCH DESIGN AND METHODS: The children will be randomly assigned to the KITS condition or a services-as-usual condition and assessed at four time points: spring prior to kindergarten, immediately prior to kindergarten entry, kindergarten fall, and kindergarten spring; 160 of the children will also be assessed in first grade spring.

MEASURES AND KEY OUTCOMES: Our multimethod, multi-informant outcome measures will include the following: direct assessments of early literacy and social-emotional skills prior to kindergarten and literacy skills and social-emotional functioning during kindergarten and first grade; parent and teacher reports on child skills and behaviors, parent involvement in early literacy and school, and parenting practices; direct classroom observations of child academic engaged time and social behaviors; and school records data on grades, office discipline referrals, special education services received, and attendance.

DATA-ANALYTIC STRATEGIES: Analyses will employ variable-centered (e.g., ANOVA and regression) and person-centered (e.g., latent growth curve modeling) approaches. Multilevel latent variable modeling will be used to test how changes in hypothesized mediators affect longer-term outcomes and how outcomes vary depending on level of hypothesized moderators.

ELIGIBILITY:
Inclusion Criteria:

* Child is entering kindergarten in a disadvantaged neighborhood
* Child is a bilingual or monolingual English speaker

Exclusion Criteria:

* Child has a hearing or vision impairment that would limit participation in the intervention activities or assessment protocol

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 265 (Actual)
Dates: Start 2013-03; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Change in early literacy skills from baseline to kindergarten fall | pre-intervention (baseline), pre-kindergarten (average of 2-3 months post baseline), kindergarten fall (average of 4-5 months post-baseline)
  Standardized measures of early literacy skills including letter naming, phonological awareness and understanding of concepts about print
Change in prosocial skills from baseline to kindergarten fall | pre-intervention (baseline), pre-kindergarten (average of 2-3 months post baseline), kindergarten fall (average of 4-5 months post-baseline)
  Standardized direct assessments of the child's responses to social situations as well as parent and teacher responses to standardized questionnaires on children's social skills
Change in emotion and behavior regulation skills from baseline to kindergarten fall | pre-intervention (baseline), pre-kindergarten (average of 2-3 months post baseline), kindergarten fall (average of 4-5 months post-baseline)
  Standardized direct assessment of the children's executive function skills as well as parent and teacher report on standardized questionnaires used to assess emotion and behavior regulation
Change in parenting behavior (parent involvement and positive parenting practices) from baseline to kindergarten fall | pre-intervention (baseline), pre-kindergarten (average of 2-3 months post baseline), kindergarten fall (average of 4-5 months post-baseline)
  Caregiver reported involvement in early literacy activities and beliefs about the importance of various literacy skills for kindergarten as well as parenting practices

SECONDARY OUTCOMES:
Longitudinal academic achievement across grade levels | post-kindergarten (average of 12 months post-baseline), post-first grade (average of 24 months post-baseline)
  Standardized direct assessments of child achievement in reading and math as well as parent and teacher report on standardized measures of child achievement.
Longitudinal social competence across grade levels | post-kindergarten (average of 12 months post-baseline), post-first grade (average of 24 months post-baseline)
  Standardized direct child assessments of responses to peer situations as well as child report on standardized questionnaires about social functioning at school and parent and teacher reports of child social functioning on standardized questionnaires
Longitudinal parenting behaviors (parental involvement and positive parenting) | post-kindergarten (average of 12 months post-baseline), post-first grade (average of 24 months post-baseline)
  Caregiver and teacher reports on parental involvement in school as well as positive parenting practices

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Pears, Ph.D., Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

REFERENCES:
- [Background] Pears KC, Kim HK, Fisher PA. Effects of a School Readiness Intervention for Children in Foster Care on Oppositional and Aggressive Behaviors in Kindergarten. Child Youth Serv Rev. 2012 Dec;34(12):2361-2366. doi: 10.1016/j.childyouth.2012.08.015. No abstract available. PMID 23710106
- [Background] Pears KC, Fisher PA, Bronz KD. An Intervention to Promote Social Emotional School Readiness in Foster Children: Preliminary Outcomes From a Pilot Study. School Psych Rev. 2007;36(4):665-673. PMID 19057655
- [Background] Pears KC, Healey CV, Fisher PA, Braun D, Gill C, Conte HM, Newman J, Ticer S. Immediate Effects of a Program to Promote School Readiness in Low-Income Children: Results of a Pilot Study. Educ Treat Children. 2014 Aug;37(3):431-460. doi: 10.1353/etc.2014.0021. PMID 25382932
- [Result] Pears KC, Fisher PA, Kim HK, Bruce J, Healey CV, Yoerger K. Immediate Effects of a School Readiness Intervention for Children in Foster Care. Early Educ Dev. 2013 Aug;24(6):771-791. doi: 10.1080/10409289.2013.736037. PMID 24015056
- [Result] Pears KC, Kim HK, Fisher PA. Decreasing Risk Factors for Later Alcohol Use and Antisocial Behaviors in Children in Foster Care by Increasing Early Promotive Factors. Child Youth Serv Rev. 2016 May;65:156-165. doi: 10.1016/j.childyouth.2016.04.005. PMID 27158175
- See also: Related Info — http://www.oslc.org